CLINICAL TRIAL: NCT05022758
Title: RENal Outcomes of Rivaroxaban Compared With Warfarin in Asian patienTs With nOn-valvular atRial Fibrillation: a Nationwide Population-based Study
Brief Title: A Study to Learn Whether There Are Differences in the Kidney's Ability to Work Properly in Korean Patients With Non-valvular Atrial Fibrillation (Irregular and Often Rapid Heartbeat Not Caused by a Heart Valve Problem) Treated With Rivaroxaban as Compared to Those Treated With Warfarin
Acronym: RENOVATOR
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 21615
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Non-valvular Atrial Fibrillation (NVAF)
Keywords: Non-valvular atrial fibrillation (NVAF); Stroke; Rivaroxaban; Systemic embolism
MeSH Terms: conditions — Stroke | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants treated with rivaroxaban: NVAF patients who were OAC-naïve (Have no record of Oral anticoagulation [OAC] therapy use in the January 2013 to December 2014) and newly initiated on rivaroxaban (defined as the index date) during the enrollment period from January 2015 to December 2017.
  Interventions: Drug: Rivaroxaban (Xarelto, BAY59-7939)
- Participants treated with warfarin: NVAF patients who were OAC-naïve (Have no record of Oral anticoagulation [OAC] therapy use in the January 2013 to December 2014) and newly initiated on warfarin (defined as the index date) during the enrollment period from January 2015 to December 2017.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban (Xarelto, BAY59-7939) — One of NOAC (Non-vitamin K antagonist oral anticoagulants)
  Groups: Participants treated with rivaroxaban
Drug: Warfarin — One of OAC (Oral anticoagulation therapy)
  Groups: Participants treated with warfarin

SUMMARY:
This is an observational study in which data collected from the past of patients with non-valvular atrial fibrillation (NVAF) is studied.

NVAF is a condition in which patients suffer from irregular and often rapid heartbeats which are not caused by a heart valve problem. NVAF can lead to thromboembolism, a condition that happens when a blood clot forms in the body and travels through the blood stream to plug another vessel. To prevent thromboembolism doctors often prescribe a blood thinner medication.

In patients with NVAF that receive a blood thinner, it is common that the kidneys' ability to work properly, also called the kidney function, decreases. This may increase the risk of stroke, a condition which occurs when a vessel supplying blood to the brain is blocked and the risk of bleeding. It is therefore important to maintain the kidneys' ability to work properly in these patients who are treated with blood thinners.

In the beginning, only one blood thinner that could be given as a tablet by mouth was available. This blood thinner was called warfarin. Over the years, further medications have become available, for example dabigatran or rivaroxaban. There is some evidence that a decrease of the kidney function is more common with warfarin than with dabigatran or rivaroxaban. For other similar new treatments however, evidence is missing or conflicting. There also could be other relevant factors such as the kidney function before the start of treatment or the patient's genes/origin.

In this study researchers want to collect more data to compare two different blood thinner medications, rivaroxaban and warfarin. The main goal is to see whether there is a difference between the two treatments regarding the kidneys' ability to work properly. To find this out, the researchers will compare the number of patients in each group who developed chronic kidney disease stage 5 (close to or corresponding to chronic kidney failure), had a kidney transplant or needed to undergo long term dialysis. In addition, data is collected and compared about the patients' age, gender, weight, height and whether they had other related medical problems.

This study will collect information from the health records from the Korean National Health Insurance Corporation (NHIC) database. Besides this data collection, no further tests or examinations are planned in this study. Researchers will look at the health information from adult men and women in Korea who were diagnosed with NVAF between January 2013 and December 2017. They will study data of the patients who did not receive any medication with blood thinners in past 24 months before starting rivaroxaban and warfarin treatment between January 2015 and December 2017. They will follow up all the participants until December 2018.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥20 years of age (legal age in Korea) at the time of anticoagulation initiation
* Have a diagnosis of NVAF (in the 24-months prior to index date)
* Have no record of OAC use (in the 24-months prior to index date)
* Newly initiated on rivaroxaban or warfarin (index date)

Exclusion Criteria:

* Who have end-stage renal disease or are on dialysis (in the 12-months prior to index date)
* With evidence of valvular heart disease (in the 12-months prior to index date)
* With pulmonary embolism or deep vein thrombosis (within 6 months before index date)
* Who received joint replacement (within 6 months before diagnosis)
* Patients who had previous OAC prescription between 2013 and 2014
* With rivaroxaban doses other than 15 or 20 mg once daily

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study is conducted using administrative claims data of the Korean National Health Insurance Service (NHIS) and the linked health check-up database of the National Health Insurance Corporation (NHIC) between 2013 to 2018.
Sampling Method: Non-Probability Sample
Enrollment: 45000 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incidence of kidney failure | Retrospective analysis from 01-Jan-2015 to 31-Dec-2018
  Kidney failure is defined as progression to stage 5 chronic kidney disease (CKD), the need for maintenance dialysis, or having a kidney transplant

SECONDARY OUTCOMES:
Number of participants with ≥ 30% decline in estimated glomerular filtration rate (eGFR) | Retrospective analysis from 01-Jan-2015 to 31-Dec-2018
Number of participants with doubling of the serum creatinine level | Retrospective analysis from 01-Jan-2015 to 31-Dec-2018
Incidence of Acute kidney injury (AKI) | Retrospective analysis from 01-Jan-2015 to 31-Dec-2018
  AKI is defined as an emergency department visit or hospitalization with a diagnostic code of AKI
Number of participants with composite renal outcome of ≥ 30% decline in eGFR, doubling of the serum creatinine level and kidney failure | Retrospective analysis from 01-Jan-2015 to 31-Dec-2018

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, South Korea

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.